CLINICAL TRIAL: NCT02990156
Title: Prospective, Randomized, Controlled, Open Label, All China, Multi-Center, Registration Trial of the MICROPORT NEUROTECH Coil Embolization System for the Traetment of Intracranial Aneurysms
Brief Title: CATCH [Short Name for: Coil Application Trial in China]
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-Nemo-01-A
Record Dates: First submitted 2016-12-01; First posted 2016-12-13 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Intracranial Aneurysm
Keywords: Coils
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coil Embolization System (Experimental): Coil Embolization System,or deposits coils in the aneurysm sac by electrolytical detachment; coil types include Complex Finish, Complex Frame,and Helical. The coils are made of a platinum - tungsten alloy, have a minimum diameter of 2 mm and a maximum diameter of 24mm.
  Interventions: Device: Coil Embolization System
- Control device from Medronic (Active Comparator): Control device from Medronic,include AxiumTM Detachable Coils and AxiumTM Prime Detachable Coils, which are manufactured by ev3 (Medtronic, Irvine, California, USA);
  Interventions: Device: Cotrol device from Medronic

INTERVENTIONS:
Device: Coil Embolization System — deposits coils in the aneurysm sac by electrolytical detachment; coil types include Complex Finish, Complex Frame, and Helical. The coils are made of a platinum - tungsten alloy, have a minimum diameter of 2 mm and a maximum diameter of 24mm. The intended use of the Microport NeuroTech Coil Embolization System is for the endovascular embolization of intracranial aneurysms.
  Arms: Coil Embolization System
Device: Cotrol device from Medronic — Control device from Medronic (include AxiumTM Detachable Coils and AxiumTM Prime Detachable Coils) are manufactured by ev3 (Medtronic, Irvine, California, USA);
  Arms: Control device from Medronic

SUMMARY:
The scope of this trial is the collection and analysis of effectiveness and safety endpoints, related to the use of the MicroPort NeuroTech Coil Embolization System in the treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
A cerebral aneurysm (also known as an intracranial or intracerebral aneurysm) is a weak or thin spot on a blood vessel in the brain that balloons out and fills and intermixes with parent artery blood. Aneurysms can occur at any age. Global incidence varies by country, with reports of prevalence ranging from 5.1 to 19.6 cases per 100,000 persons. With the development of imaging technology and the greater attention paid by people to their overall health,there will be more aneurysms be detected. The combination of sophisticated imaging equipment, more frequent use of imaging in patients, and the aforementioned emphasis on optimum health, has led to a greater proportion of asymptomatic aneurysms being discovered.

The most common type of aneurysms are saccular; and, aneurysms are more likely to occur in women. The most devastating presentation of an intracranial aneurysm is subarachnoid hemorrhage (SAH). It is estimated that, on average, five percent of the population is afflicted and the incidence of aneurysm rupture (SAH) is between 6 and 9 per 1000 000 individuals . Mortality can approach 50%, with fewer than 60% of survivors returning to independent living.

Invasive treatment of aneurysms began with an open surgical procedure referred to as 'surgical clipping'. This treatment was once considered the gold standard treatment for aneurysms. The first neurovascular interventional medical device was the Guglielmi Detachable Coil (GDC), which was developed and tested in the mid-1990s and was introduced by Dr. Guido Guglielmi and Target Therapeutics, Fremont, California. These bare platinum coils were electrolytically detached for placement in the aneurysm sac. It took approximately one decade to prove coiling superiority over surgical clipping, after publication of the results of the ISAT Study. Since that time, coils have become more sophisticated in makeup and conformation. Coil use is also a mainstay for neurovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old and ≤80 years old at the time of signing the informed consent;
2. Intracranial ruptured or unruptured, single, previously untreated, saccular aneurysm diagnosed by CTA, MRA, DSA or other similar neuroimaging examination;
3. The maximum diameter of target aneurysm ≤24mm;
4. Baseline modified Rankin score (mRS) ≤2 points;
5. Baseline Hunt - Hess scores of patients with ruptured aneurysm ≤ Ⅲ;
6. The target aneurysm can be embolized in one operation;
7. The patient or the patient's guardian signs the informed consent voluntarily and is willing to accept follow-up.

Exclusion Criteria:

1. Clear allergy, resistance or contraindication to antiplatelet drugs, anticoagulants, contrast agents and/or anesthetics.
2. Definite allergy to platinum, tungsten and/or any substances of coils.
3. Subjects who are not suitable for anesthesia or endovascular treatment, such as those suffering from severe respiratory system, liver and kidney diseases or coagulation disorders (such as hemophilia).
4. Target aneurysm parent vessel stenosis ≥70%.
5. Anatomy not appropriate for endovascular treatment due to severe intracranial vessel tortuosity or stenosis, or intracranial vasospasm not responsive to medical therapy.
6. The target aneurysm has previously received surgery or other endovascular treatment.
7. Ruptured aneurysm requiring stent-assisted embolization.
8. The target aneurysm is hemangioid aneurysm, dissected aneurysm, fusiform aneurysm, infectious aneurysm, pseudoaneurysm, or arteriovenous malformation, or aneurysm associated with Moyamoya disease.
9. Major surgery was performed within 30 days before enrollment, or surgery was planned within 90 days after enrollment.
10. Patients with active infection at puncture point or other serious infection are not suitable for endovascular treatment.
11. Illness with a potential risk of sudden death.
12. Subjects with intracranial space-occupying lesions (e.g., intracranial tumor, abscess, etc.) or who are receiving radiotherapy for their head and neck.
13. Long-term treatment with anticoagulant drugs (such as warfarin) is required.
14. Having cognitive impairment, psychiatric disorder or other medical condition that may affect the data evaluation or trial results.
15. Unable to understand the trial or has a record of noncompliance with medical advice.
16. Taking banned medicine.
17. Life expectancy less than 1 year, may not complete follow-up.
18. Women in pregnancy or lactation, or women with positive pregnancy test.
19. Subjects who are participating in clinical trials of other drugs or devices and have not reached the end point of the trial, or are expected to participate in clinical trials of other drugs or devices.
20. Investigators do not consider it appropriate to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Raymond Scale | 6 Months
  For the MicroPort NeuroTech Coil Embolization System, this endpoint will be based upon the 6-month Core Lab identification of patients with "Successful occlusion" rate: % of subjects who at 6 months' post coiling, reported as a combination of Raymond 1 and Raymond 2 outcomes (95%-100%). The endpoint will be expressed as a percentage of all evaluable subjects with complete and nearly complete (95%-100%) occlusion in the context of the whole population of evaluable subjects (n/N).

SECONDARY OUTCOMES:
Modified Rankin Scale | 6 Months
  6-months post-treatment "Clinical Worsening", "Clinical Worsening" will be calculated as the percentage of subjects who meet the following condition: Final mRS score is more than 2 and is at least 1 point higher than the pre study measurement.
  For most subjects, this will be determined at the 6-months follow up visit. However, for those subjects whose trial participation is prematurely shortened, as a result of death (mRS will count as 6) or very serious device or procedure related debilitating injury, their final mRS determination will be counted, as the most recent score at the time of leaving the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin LIU, MD, Principal Investigator — Changhai Hospital
Locations (1):
- MicroportNT, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jin Y, Guo X, Quan T, Zhao R, Li T, Zhao Z, Yang H, Zhu X, Liang G, Leng B, Wu X, Wang Y, Guan S. Randomized, prospective, multicenter trial assessing the numen coil embolization system in the endovascular treatment of small intracranial aneurysms: outcomes from the CATCH Trial. BMC Surg. 2023 Jun 16;23(1):164. doi: 10.1186/s12893-023-02049-9. PMID 37328839